CLINICAL TRIAL: NCT06390319
Title: SJALL23T: Adding Dasatinib Or Venetoclax To Improve Responses In Children With Newly Diagnosed T-Cell Acute Lymphoblastic Leukemia (ALL) Or Lymphoma (T-LLY) Or Mixed Phenotype Acute Leukemia (MPAL)
Brief Title: Adding Dasatinib Or Venetoclax To Improve Responses In Children With Newly Diagnosed T-Cell Acute Lymphoblastic Leukemia (ALL) Or Lymphoma (T-LLY) Or Mixed Phenotype Acute Leukemia (MPAL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJALL23T; NCI-2024-03015 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; T-cell Lymphoma; Mixed Phenotype Acute Leukemia
Keywords: Newly Diagnosed; Children; Young Adults; T-cell Acute Lymphoblastic Leukemia; T-cell Lymphoma; Mixed Phenotype Acute Leukemia (MPAL)
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell; Leukemia, Biphenotypic, Acute | interventions — Dexamethasone; Calcium Dobesilate; Vincristine; Daunorubicin; calaspargase pegol; Dasatinib; venetoclax; Bortezomib; Methotrexate; Hydrocortisone; Cytarabine; Cyclophosphamide; Mercaptopurine; nelarabine; Thioguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Patients with T-ALL (except ETP or near-ETP) (Experimental): All eligible patients receive intervention according to the Detailed Description section with the following:
  Induction: Dexamethasone, Vincristine, Daunorubicin, Calaspargase pegol, Dasatinib, IT MHA
  Early Post Induction: Cyclophosphamide, Cytarabine, Mercaptopurine, Nelarabine, IT MHA, Methotrexate, Dasatinib, Dexamethasone, Vincristine, Daunorubicin, Calaspargase pegol
  Maintenance: Mercaptopurine, Methotrexate, Nelarabine, Cyclophosphamide, Cytarabine, Dexamethasone, Vincristine, Dasatinib, IT MHA, Thioguanine
  Interventions: Drug: Dexamethasone; Drug: Vincristine; Drug: Daunorubicin; Drug: Calaspargase pegol; Drug: Dasatinib; Drug: Intrathecal triple therapy (methotrexate + hydrocortisone + cytarabine); Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Nelarabine; Drug: Methotrexate; Drug: Thioguanine
- Patients with ETP or near-ETP ALL or MPAL (Experimental): All eligible patients receive intervention according to the Detailed Description section with the following:
  Induction: Dexamethasone, Vincristine, Daunorubicin, Calaspargase pegol, Venetoclax, IT MHA
  Early Post Induction: Cyclophosphamide, Cytarabine, Mercaptopurine, Nelarabine, IT MHA, Methotrexate, Dexamethasone, Vincristine, Daunorubicin, Calaspargase pegol, Venetoclax
  Maintenance: Mercaptopurine, Methotrexate, Nelarabine, Cyclophosphamide, Cytarabine, Dexamethasone, Vincristine, IT MHA, Thioguanine
  Interventions: Drug: Dexamethasone; Drug: Vincristine; Drug: Daunorubicin; Drug: Calaspargase pegol; Drug: Venetoclax; Drug: Intrathecal triple therapy (methotrexate + hydrocortisone + cytarabine); Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Nelarabine; Drug: Methotrexate; Drug: Thioguanine
- Patients with T-LLy (Experimental): All eligible patients receive intervention according to the Detailed Description section with the following:
  Induction: Dexamethasone, Vincristine, Daunorubicin, Calaspargase pegol, Bortezomib, IT MHA
  Early Post Induction: Cyclophosphamide, Cytarabine, Mercaptopurine, IT MHA, Methotrexate, Dexamethasone, Vincristine, Daunorubicin, Calaspargase pegol, Bortezomib
  Maintenance: Mercaptopurine, Methotrexate, Cyclophosphamide, Cytarabine, Dexamethasone, Vincristine, IT MHA, Thioguanine
  Interventions: Drug: Dexamethasone; Drug: Vincristine; Drug: Daunorubicin; Drug: Calaspargase pegol; Drug: Bortezomib; Drug: Intrathecal triple therapy (methotrexate + hydrocortisone + cytarabine); Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Thioguanine

INTERVENTIONS:
Drug: Dexamethasone — Given orally (PO) or intravenously (IV).
  Other Names: Decadron; Hexadrol®
Drug: Vincristine — Given IV.
  Other Names: Vincristine Sulfate; Oncovin
Drug: Daunorubicin — Given IV.
  Other Names: Daunomycin
Drug: Calaspargase pegol — Given IV.
  Other Names: ASPARLAS
Drug: Dasatinib — Given PO
  Other Names: Sprycel®
  Arms: Patients with T-ALL (except ETP or near-ETP)
Drug: Venetoclax — Given PO (ETP, near-ETP, and MPAL only).
  Other Names: Venclexta®
  Arms: Patients with ETP or near-ETP ALL or MPAL
Drug: Bortezomib — Given IV (T-LLy only).
  Other Names: Velcade®
  Arms: Patients with T-LLy
Drug: Intrathecal triple therapy (methotrexate + hydrocortisone + cytarabine) — Given Intrathecal (IT), Age adjusted.
  Other Names: IT MHA
Drug: Cyclophosphamide — Given IV.
  Other Names: Cytoxan®
Drug: Cytarabine — Given IV or IT.
  Other Names: Ara-C; Cytosine arabinoside
Drug: Mercaptopurine — Given PO.
  Other Names: 6-MP
Drug: Nelarabine — Given IV
  Other Names: Arranon; Atriance
  Arms: Patients with ETP or near-ETP ALL or MPAL; Patients with T-ALL (except ETP or near-ETP)
Drug: Methotrexate — Given IT, IV, PO or intramuscular (IM).
  Other Names: Trexall®
Drug: Thioguanine — Given PO (participants intolerant to mercaptopurine).
  Other Names: 6-thioguanine; Tabloid®

SUMMARY:
This is a clinical trial testing whether the addition of one of two chemotherapy agents, dasatinib or venetoclax, can improve outcomes for children and young adults with newly diagnosed T-cell acute lymphoblastic leukemia and lymphoma or mixed phenotype acute leukemia.

Primary Objective

* To evaluate if the end of induction MRD-negative rate is higher in patients with T-ALL treated with dasatinib compared to similar patients treated with 4-drug induction on AALL1231.
* To evaluate if the end of induction MRD-negative rate is higher in patients with ETP or near-ETP ALL treated with venetoclax compared to similar patients treated with 4-drug induction on AALL1231.

Secondary Objectives

* To assess the event free and overall survival of patients treated with this therapy.
* To compare grade 4 toxicities, event-free survival (EFS) and overall survival (OS) of patients treated with this therapy in induction and reinduction to toxicities of similar patients treated on TOT17.

DETAILED DESCRIPTION:
Patients will be identified in the first 3 days of therapy during their treatment on INITIALL.

Treatment will consist of 3 main phases: Induction, Early Post Induction [including Consolidation, High-Dose Methotrexate, Intensification, Interim 1, Reinduction 1, Interim 2, and Reinduction 2], and Maintenance.

Induction:

* Remission Induction includes 3 days of therapy on the INITIALL classification protocol as well as the remainder of a total of 4 weeks of induction treatment on this trial. Treatment includes a total of 28 days of dexamethasone, 4 weekly doses of vincristine, 3 doses of daunorubicin, 1 dose of Calaspargase pegol, 6 doses of Intrathecal triple therapy (IT MHA), and one of 3 additional drugs. Patients with T-ALL without near-ETP or ETP phenotype (hereafter referred to simply as T-ALL) will receive 25 days of dasatinib. Patients with ETP or near-ETP ALL as well as those with MPAL will receive 14 days of venetoclax. Patients with T-LLy will receive bortezomib. Patients will have a week without chemotherapy at the end of Induction, although patients with Induction failure (MRD ≥5% disease) will proceed directly to consolidation.

Early Post Induction:

* Consolidation will be given following completion of Remission Induction Therapy. Patients will receive 2 cycles of BFM-1b therapy (a single dose of cyclophosphamide at the start of week 1, 4 daily doses of cytarabine in two consecutive weeks, and 2 weeks of mercaptopurine) separated by a week of nelarabine. Patients will have a week without chemotherapy at the end of Consolidation.
* High-dose Methotrexate will be given for 4 cycles to all patients. Patients will also receive an intrathecal chemotherapy treatment with each of the 2-week cycles and will take oral mercaptopurine continuously if tolerated.
* Intensification will be given to patients with T-ALL or ETP/ near-ETP. This therapy includes a week of nelarabine, one week of combination cyclophosphamide and cytarabine, and 1 week of rest without chemotherapy.
* Interim Therapy 1 includes 6 weeks of oral mercaptopurine, 2 weeks (5 days of each week) of dexamethasone, and two doses (weeks 1 and 4) of daunorubicin, vincristine, and calaspargase pegol.
* Reinduction Therapy 1 will consist of 3 weekly doses of vincristine, 1 dose of daunorubicin and calaspargase pegol at the start of the first week, and dexamethasone for 7 days in the first and third weeks. Patients will also receive the same additional agent received during induction based on immunophenotype.
* Interim Therapy 2 includes 6 weeks of oral mercaptopurine, two doses (weeks 1 and 4) of daunorubicin, vincristine, and calaspargase pegol.
* Reinduction Therapy 2 will consist of 3 weekly doses of vincristine, 1 dose of daunorubicin and calaspargase pegol at the start of the first week, and dexamethasone for 7 days in the first and third weeks. Patients will also receive the same additional agent received during induction based on immunophenotype.

Maintenance therapy:

* Early Maintenance Therapy follows Reinduction 2 and lasts 31 weeks. Patients will receive mercaptopurine and methotrexate interrupted by 1 week of nelarabine (week 3), 5 cyclophosphamide/ cytarabine pulses, and every 4-week dexamethasone/ vincristine pulses. For the first 32 weeks, patients will also receive every 4-week pulses including 5 days of dexamethasone and 1 dose of vincristine. Patients will receive low-dose methotrexate in all weeks when they do not receive dexamethasone or vincristine. All patients will receive every 4-week intrathecal chemotherapy beginning 4 weeks after the week of nelarabine.
* Late Maintenance Therapy follows early maintenance and includes daily mercaptopurine, weekly methotrexate, and every 8-week intrathecal chemotherapy. It lasts a total of 44 weeks.

Duration of therapy is approximately 2¼ years. It is recommended that patients be followed every 4 months for 1 year, every 6 months for 1 year and then yearly until the patient is in remission for 10 years and is at least 18 years old.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment on INITIALL.
* Age 1-18.99 years at the time of enrollment on INITIALL.
* T-Acute lymphoblastic leukemia or lymphoblastic lymphoma or mixed phenotype acute leukemia/ lymphoma
* No prior chemotherapy excluding therapy given on or allowed by INITIALL.
* Patient has completed no more than 3 days of chemotherapy on INITIALL.
* Direct bilirubin ≤ 1.5x the upper limit of normal for age
* Alanine aminotransferase (ALT) ≤ 5x the upper limit of normal for age
* Calculated glomerular filtration rate (GFR) ≥ 50 mL/min/1.73m^2 using the Bedside Schwartz equation OR creatinine below or equal to the maximum defined below:

  * Age: 1 to < 2 years - Maximum serum creatinine (mg/dL): 0.6 (Male), 0.6 (Female)
  * Age: 2 to < 6 years - Maximum serum creatinine (mg/dL): 0.8 (Male), 0.8 (Female)
  * Age: 6 to < 10 years - Maximum serum creatinine (mg/dL): 1 (Male), 1 (Female)
  * Age: 10 to < 13 years - Maximum serum creatinine (mg/dL): 1.2 (Male), 1.2 (Female)
  * Age: 13 to < 16 years - - Maximum serum creatinine (mg/dL): 1.5 (Male), 1.4 (Female)
  * Age: ≥ 16 years - Maximum serum creatinine (mg/dL): 1.7 (Male), 1.4 (Female)

Exclusion Criteria:

* Inability or unwillingness to give informed consent/ assent as applicable.
* Patients with > Grade 2 neuropathy at the time of enrollment (participant with T-LLy only).
* Documented malabsorption syndrome or any other condition that precludes receipt of oral medications.
* Known HIV infection or active hepatitis B (defined as hepatitis B surface antigen-positive) or C (defined as hepatitis C antibody-positive).
* Pregnant or lactating.
* For patients of reproductive potential, unwillingness to use highly effective contraception for the duration of protocol therapy and for 90 days afterwards.
* Receipt of a strong or moderate CYP3A4 inducer such as rifampin, carbamazepine, phenytoin, and St. John's wort within 7 days of the start of protocol treatment.
* Consumption of grapefruit, grapefruit products, Seville oranges, or starfruit within 3 days of the start of protocol therapy.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD)-negativity rate in patients with T cell acute lymphoblastic leukemia | Up to end of induction day 29 or death
  Comparison of the probability of achieving negative MRD (<0.01%) and M1 bone marrow status at the end of induction between this protocol and COG AALL1231 will be performed. Statistical analysis of the primary objective will be conducted according to a group sequential design with 1 interim analysis, by a slightly modified version of the procedure for binary endpoint.
MRD-negativity rate in patients with ETP or near ETP ALL | Up to end of induction day 29 or death
  The proportion of patients with ETP or near-ETP treated with venetoclax based induction will be compared to the rate of such unsuccessful induction in patients treated on AALL1231 with a standard 4-drug induction. The probability of achieving negative MRD will be tested using a one-sided exact binomial proportion test.

SECONDARY OUTCOMES:
Event-free survival (EFS) | Up to 10 years
  Kaplan-Meier estimates for EFS will be calculated along with standard error.
Overall survival (OS) | Up to 10 years
  Kaplan-Meier estimates for OS will be calculated along with standard error.
Incidence of grade 4 toxicities | Up to 30 days after last dose of study treatment
  Adverse events will be graded using Common Terminology Criteria for Adverse Events version 5 and compared using Fisher's or exact Chi-square test.
EFS compared to Total 17 (TOT17-NCT03117751) | Up to 10 years
  Comparisons of EFS to the corresponding TOT17 will be performed by the log-rank test.
OS compared to TOT17 | Up to 10 years
  Comparisons of OS to the corresponding TOT17 will be performed by the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Seth E. Karol, MD, MSCI, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - Rady Children's Hospital, San Diego, California
  - Saint Francis Children's Hospital, Tulsa, Oklahoma
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols